CLINICAL TRIAL: NCT00652015
Title: Molecular and Cellular Mechanisms of the In-stent-thrombosis. Is it Possible to Predict a In-stent-thrombosis Using Biomarkers?
Brief Title: Molecular and Cellular Mechanisms of the In-stent-thrombosis
Status: Withdrawn | Type: Observational
Why Stopped: Recruitment numbers could not at all been achieved in an acceptable period of time
Sponsor: RWTH Aachen University (Other)
Responsible Party: Burcin Özüyaman, MD, RWTH Aachen University
Other Study IDs: EK 039/08
Record Dates: First submitted 2008-03-31; First posted 2008-04-03 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Patients With SAT or LT After Stent Implantation (PCI)
Keywords: in-stent-thrombosis; CD39; CD73; EPC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1 sample of approximately 30 mL blood will be taken from each patient of both study group.
  CD39 and CD73 activity as well as EPC-number and function will be analyzed.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients having developed an in-stent-thrombosis (40 SAT, 40 LT)
- 2: Patients having not developed an in-stent-thrombosis after stent implantation using PTCA

SUMMARY:
In-Stent-Thrombosis is a rare but serious complication after implantation of stents during PTCA.

DETAILED DESCRIPTION:
In this prospective, open, not-randomized, controlled single-center pilot study 80 patients having had an in-stent-thrombosis (40 sub-acute thromboses (SAT), 40 late thromboses (LT)) and a control group of 80 patients having not developed a thrombosis will be compared.

The aim of this study is the establishment of diagnostic markers vor prediction of SAT (detection of CD39- and CD73-activity, respectively)and of LT (EPC-number and function, respectively) correspondingly aiming at the early identification of patients with high risk for developing an in-stent-thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* patients having developed an SAT or LT after stent implantation using PTCA

Exclusion Criteria:

* instabel coronary heart diseases,
* systemic autoimmune diseases,
* rheumatic diseases,
* tumors,
* impaired kidney or liver function,
* surgery within the last 3 months,
* pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients having developed an SAT or LT after stent implantation using PTCA
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
The aim of this study is to establish diagnostic markers for prediction of SAT and LT, respectively, by identification of CD39 and CD73-activity and EPC-number and function, respectively. | may 08 to may 2010

CONTACTS AND LOCATIONS:
Overall Officials: Burcin Özüyaman, MD, Principal Investigator — RWTH Aachen University
Locations (1):
- RWTH University Hospital, Aachen, Germany